CLINICAL TRIAL: NCT00943592
Title: Clofarabine-melphalan-alemtuzumab Conditioning in Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14341B; NCT00572546 (obsolete NCT alias)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Hematologic Malignancies; Leukemia; Preleukemia
Keywords: Melphalan; Alemtuzumab; Clofarabine
MeSH Terms: conditions — Leukemia; Preleukemia | interventions — Clofarabine; Melphalan; Alemtuzumab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Clofarabine; Drug: Melphalan; Drug: Campath; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Clofarabine — Clofarabine will be administered as a 2-hour IV infusion on Days 1 through 5 at approximately the same time everyday (4 dose levels).
Drug: Melphalan — Doses ranging from 100 to 140 mg/m2
Drug: Campath — 20mg/d x5
Procedure: Stem Cell Transplant — Infusion of donor, bone marrow and auto.

SUMMARY:
This is a clinical research study designed to evaluate whether a conditioning regimen consisting of the combination of three drugs named melphalan, alemtuzumab and clofarabine supported by donor blood cells will result in rapid recovery and a high rate of long-lasting remissions in patients with leukemia, lymphoma and myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute myelogenous or lymphoid leukemia
* Chronic myelogenous leukemia in accelerated phase or blast-crisis
* Chronic myelogenous leukemia in second or subsequent chronic phase
* Recurrent or refractory malignant lymphoma or Hodgkin's disease
* Multiple myeloma at high risk for disease recurrence
* Chronic lymphocytic leukemia, relapsed or with poor prognostic features
* Other Myeloproliferative disorder (polycythemia vera, essential thrombocythemia, myelofibrosis) with poor prognostic features
* Myelodysplastic syndromes (including PNH) with > 5% blasts
* Zubroid performance status < 2 (See Appendix B)
* Life expectancy is not severely limited by concomitant illness
* Adequate cardiac and pulmonary function. Patients with decreased LVEF or PFTS will be evaluated by cardiology or pulmonary prior to enrollment on this protocol
* Calculated Creatinine Clearance > 50 ml/min
* Serum bilirubin 2.0 mg/dl, SGPT < 3x upper limit of normal
* No evidence of chronic active hepatitis or cirrhosis
* HIV-negative
* Patient is not pregnant
* Patient or guardian able to sign informed consent

Exclusion Criteria:

* Clinical progression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2006-03; Primary Completion 2011-04 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine, Melphalan, and Alemtuzumab: Clofarabine was initially administered IV infusion over 1 hour on days -7 through -3 (4 dose levels from 10 to 40 mg/m2); subsequently, the protocol was amended to infuse clofarabine over 3 hours. Melphalan (doses ranging from 100 to 140 mg/m2) was infused over 30 minutes on day -2. Alemtuzumab was administered at 20 mg IV infusion on day -7 through day -3 over 1 hour.
Period: Overall Study
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Started | 82
Maximum Tolerated Dose | 74 (74 patients received the Maximum Tolerated Dose)
Completed | 79 (None of the three deaths were attributed to the conditioning regimen)
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 82
Age, Continuous [Median (Full Range); unit: years] | 54 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hepatic Adverse Events During the Conditioning Regimen Prior to Stem Cell Transplantation
Description: Toxicity was scored according to NCI/CTC version 3
Time Frame: Day 7 until Day 30
Measure: Number; unit: participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 82
participants
  Grade 1-2 | 48
  Grade 3-4 | 30

2. Secondary Outcome: Overall Survival (OS)
Time Frame: 1 year
Population: 74 patients received the Maximum Tolerated Dose of clofarabine 40 mg/m2 IV daily x 5 days, melphalan 140 mg/m2 x 1 day, and alemtuzumab 20 mg IV daily x 5 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 74
percentage of participants | 59 [47 to 71]

3. Primary Outcome: Number of Participants With Renal Adverse Events During the Conditioning Regimen Prior to Stem Cell Transplantation
Description: Toxicity was scored according to NCI/CTC version 3
Time Frame: Day 7 until Day 30
Measure: Number; unit: participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 82
participants
  Grade 1-2 | 26
  Grade 3-4 | 13
  Grade 5 | 3

4. Primary Outcome: Number of Participants With Skin Adverse Events During the Conditioning Regimen Prior to Stem Cell Transplantation
Description: Toxicity was scored according to NCI/CTC version 3
Time Frame: Day 7 until Day 30
Measure: Number; unit: participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 82
participants
  Grade 1-2 | 6
  Grade 3-4 | 8

5. Primary Outcome: Number of Participants With Other Adverse Events During the Conditioning Regimen Prior to Stem Cell Transplantation
Description: Toxicity was scored according to NCI/CTC version 3
Time Frame: Day 7 until Day 30
Measure: Number; unit: participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 82
participants
  Grade 1-2 | 12
  Grade 3-4 | 7
  Grade 5 | 7

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression is defined from stem cell infusion to disease relapse, i.e., recurrence of hematologic malignancy and/or need for treatment after transplant for disease or death from any cause, whichever occurred first.
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 74
percentage of participants | 45 [33 to 67]

7. Secondary Outcome: Treatment-related Mortality (TRM)
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 74
percentage of participants | 26 [16 to 36]

8. Secondary Outcome: Relapse Rate
Time Frame: 1 year
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Number analyzed (Participants) | 74
percentage of participants | 29 [18 to 40]

ADVERSE EVENTS:
Arm/Group | Clofarabine, Melphalan, and Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 44/82
Other Adverse Events (participants affected / at risk) | 62/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Melphalan, and Alemtuzumab (N=82)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiovascular disease, unspecified (Cardiac disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4)
Mucositis (General disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (8)
Renal disorder NOS (Renal and urinary disorders) | 16 (16)
Hepatobiliary disease NOS (Hepatobiliary disorders) | 30 (30)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Melphalan, and Alemtuzumab (N=82)
Anxiety (Psychiatric disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Hepatobiliary disease NOS (Hepatobiliary disorders) | 48 (48)
Mucositis (General disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Renal disorder NOS (Renal and urinary disorders) | 26 (26)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pseudotumor cerebri (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No